CLINICAL TRIAL: NCT05935488
Title: Breath Detection of Non-alcoholic Steatohepatitis (NASH)-Induced Metabolic Alterations Using Food Flavors.
Brief Title: Early Liver Disease Breath Detection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Owlstone Ltd (Industry)
Collaborators: North Norfolk Primary Care Practices (Unknown); Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other)
Responsible Party: Sponsor
Other Study IDs: OML-004
Record Dates: First submitted 2023-06-16; First posted 2023-07-07 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2023-10

CONDITIONS: Liver Fibrosis; NASH; Liver Diseases
MeSH Terms: conditions — Liver Cirrhosis; Liver Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early Liver Disease: A total of 30 subjects with fibroscan confirmed liver fibrosis likely due to non-alcoholic steatohepatitis (NASH) will be recruited.
  Interventions: Other: EVOCs emulsion

INTERVENTIONS:
Other: EVOCs emulsion — Continuous breath sampling directly into SIFT-MS equipment. The instrument is equipped with a mouthpiece connected to the SIFT inlet where the subject blows in and the breath is analyzed in real-time
  Other Names: Selected-ion flow-tube mass spectrometry (SIFT-MS)

SUMMARY:
The Early Liver Disease Breath Detection Study is a cross-sectional study where subjects with advanced liver fibrosis will ingest a mixture of food-grade compounds (known as Exogenous Volatile Organic Compound or EVOCs) in the form of an emulsion and then provide multiple breath samples. These EVOCs can be measured on exhaled breath and it has been found that liver diseases can affect the way EVOCs are processed in the body. The objective is to identify if changes in the way these EVOCs are processed in the body can have the potential to diagnose early stage liver diseases for these subjects. Subjects with fibro-scan confirmed fibrosis will be recruited from Norfolk and Norwich University Hospital (NNUH) by local research staff, they will be invited to take part in the study at a dedicated clinic at OneNorwich Practises a clinic based in Norwich City Centre. They will be asked to fast overnight then provide a baseline breath sample, before ingesting the food-grade EVOCs emulsion and then providing additional breath samples at subsequent time points up to 90 minutes post ingestion.

DETAILED DESCRIPTION:
The diagnosis of non-alcoholic steatohepatitis (NASH) still requires liver biopsy, an invasive procedure that can lead to complications. Impaired hepatic function, associated with chronic liver diseases, changes the metabolic pathways responsible for the biotransformation of certain volatile organic compounds (VOCs) exhaled in breath. Consequently, abundance of these VOCs on breath changes in the presence of chronic liver diseases and could be used as a non-invasive diagnostic tool. To date, identified VOCs with classification performance for chronic liver diseases are of exogenous origin and their abundance on breath is not only related to liver malfunction, but also to the extent of the everyday exposure to these compounds, mainly through dietary intake. To overcome this limitation, we established the exogenous volatile organic compound (EVOC) approach, based on the administration of a defined dose of a compound followed by its measurement on breath at different timepoints. We tested several compounds in healthy subjects and found that their levels on breath peak ~10 minutes after administration, followed by a progressive reduction. NASH-associated alterations of gene expression [1], and/or impaired hepatic function is expected to alter the reduction of administered compound on breath allowing for classification between NASH subjects and healthy controls. We plan to administer a cocktail of EVOCs made of limonene, benzyl alcohol, 2- pentanone, 2-butanol, and nonanal, compounds safe for human consumption, approved, and widely used in the European Union as food flavoring agents. The amounts we will administer are well below thresholds found to cause side effects in human or animal models. The working hypothesis is that NASH-induced changes of hepatic clearance of administered food flavors alters their amounts measured in breath allowing differentiation between NASH and healthy liver conditions. We aim to conduct a cross-sectional study with the objective to identify if changes in EVOCs metabolism have a diagnostic potential for subjects with advanced fibrosis.

Subjects with FibroScan-confirmed fibrosis are asked to fast overnight. Then they provide a baseline breath sample, followed by oral administration of the EVOCs cocktail, and sampling of additional breath samples at subsequent timepoints up to 90 minutes post ingestion

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent.
* >18 years old.
* Body weight > 50 kg.
* Alcohol consumption - does not drink to excess (>30 g/day in men, >20 g/day in women).
* Fibroscan kilopascal (kPa) between 8.5 and 13.5 within 6 months and/or a liver biopsy within the last 3 years showing a fibrosis activity score ≥ F2 and a NAS score > 4 with a diagnosis of non alcoholic steatohepatitis (NASH)

Exclusion Criteria:

* (Anticipated) inability to complete the breath sampling procedure due to e.g. inability to maintain adequate ventilation unaided or claustrophobia / Inability to comply with the study procedures in the opinion of the investigator.
* Participant has cirrhosis.
* Participant has current hepatocellular carcinoma (HCC) or currently being treated for HCC. Those previously with/treated for and now clear of HCC can be recruited.
* Participant's cause of liver disease is known to be one of alcohol abuse, hepatitis, autoimmune hepatitis, medications, haemochromatosis, alpha1 antitrypsin deficiency, Wilson disease, biliary problems.
* Presence of current common cold or any other infectious disease including any recent symptoms of Covid-19.
* Participant is known to be pregnant or breast feeding.
* Participant with a diagnosis of chronic, active gastritis
* Participant is affected by asthma, chronic obstructive pulmonary disease (COPD), and/or airway hyperactivity.
* Known intolerances and/or allergies (*) to any food containing tested compounds. For limonene, citrus fruits, and fruit juices. For benzyl alcohol, apricots, cranberries, and cocoa. For 2-pentanone cheddar cheese, ripe bananas, and defatted soybean flour. For 2-butanol cheddar cheese and yogurt. For nonanal, apple, avocado, black currants, cooked beef, cucumber, fish, grapefruit, lemon, lime, mandarin, orange, and peach.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 30 subjects with fibroscan confirmed liver fibrosis likely due to NASH will be recruited. To be eligible for the study participation, subjects must meet the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the potential of using breath profiles of administered flavoring compounds and their metabolites to assess liver fibrosis. | Through study completion, an average of 4 months
  To determine this the breath profiles of subjects with liver fibrosis will be compared to the breath profiles from a previously measured healthy cohort.

SECONDARY OUTCOMES:
To demonstrate intra-subject variability in NASH patients is comparable to that in healthy volunteers observed previously. | Through study completion, an average of 4 months
To demonstrate that there are correlations between abundance of EVOCs and/or their metabolites on breath and fibrosis stage and scoring determined by blood metrics or imaging modalities previously collected. | Through study completion, an average of 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- North Norfolk Primary Care, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No